CLINICAL TRIAL: NCT03949647
Title: Collection of Bone Marrow Aspirate From Normal Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919090; 19-AG-N090
Record Dates: First submitted 2019-05-11; First posted 2019-05-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01-12

CONDITIONS: Normal Aging
Keywords: LGR; Aging; CD44; Stem Cells; Progenitor Cells; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy males and females aged 18 years and older

SUMMARY:
Background:

Bone marrow is the soft material found inside most large bones of the body. Bone marrow produces red blood cells, white blood cells, and platelets that are released into the blood stream. Inside the marrow, these cells start off as young, immature cells called progenitor cells. Researchers want to study these cells in healthy people.

Objective:

To understand how progenitor cells change with age.

Eligibility:

Healthy people ages 18 and older

Design:

Participants will be screened with a questionnaire, a physical exam, and blood tests.

Participants will have a bone marrow aspirate. They will be asked to lie on their stomach or side. A local anesthetic will be injected with a small needle under the skin at the site. A needle will then be placed through the skin and into the hip bone. A small amount of the liquid part of the bone marrow will be taken up into the needle. After the needle is removed, a pressure bandage will be placed on the site.

Participants will be asked to become a repeat volunteer and have a bone marrow aspirate sample collected once every other year. They will have a physical exam and blood tests before each collection.

The cells from the collection will be used for genetic testing and research.

Participants will be in the study for as long as they remain healthy and willing to participate.

DETAILED DESCRIPTION:
Bone marrow is soft tissue found inside the large bones of the body. Bone marrow produces red blood cells, white blood cells, and platelets that are eventually released into the blood stream. These three cell types are considered mature cells (adult cells) and they come from a progenitor cell that lives in the bone marrow. This study is designed to provide bone marrow aspirate and blood cells for research studies by basic investigators within NIA. Volunteers are screened by a health history questionnaire, a physical examination by the principal investigator, and blood tests to detect any obvious blood diseases, or bleeding or immune disorders. A bone marrow aspirate procedure is performed using a needle inserted into the hip bone to withdraw a small amount of fluid from the bone marrow for studies. NIA Researchers will use these samples for in vitro research only. In other words, these cells are never given back to a human. We will not share samples or data with researchers outside NIH.

The study population consists of healthy males and females aged 18 years and older. Study subjects are anticipated to be non-patient community volunteers. Individuals will not be excluded based on gender, race, or ethnicity. The number of subjects to be enrolled will be 2000. This will allow us to try and maintain 200 active participants in this protocol. Volunteers are screened initially and once every 2 years while on-study by a health history questionnaire and laboratory testing. Although participants may undergo a bone marrow aspirate procedure every 56 days in clinical practice, it is our plan to collect longitudinal data and obtain one sample once every other year.

We will collect bone marrow aspirate samples for distribution to NIA research investigators for their studies of the aging process in progenitor cells. We will be performing bone marrow aspirate collections of 1-5 samples every other week. We will need to maintain an active volunteer pool of approximately 200 active volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Normal healthy males and females, age 18 years and older.
  2. Agree to DNA/RNA extraction of collected samples, and analysis and storage.
  3. Health History Questionnaire, based on the American Association of Blood Banks (AABB) guidelines (Attachment 3), is not remarkable for active infection or HIV risk.
  4. Able to speak and read English.
  5. Willingness and ability to come to the NIA Clinical Research Unit at MedStar Harbor Hospital in Baltimore every 2 years for a bone marrow aspiration procedure.

EXCLUSION CRITERIA:

1. Unable to verify identification of volunteer by state issued ID card, driver s license, or military ID. Participants earning greater than $600.00/year are issued a 1099 form, therefore, positive identification is required.
2. Unable to provide informed consent
3. Allergy to Lidocaine (numbing agent) used during bone marrow aspiration procedure
4. Test results are positive for viral infections such as RPR, HIV, Hepatitis B surface antigen or hepatitis C antibodies. For participants who have been treated for Hepatitis C, screening blood work must show HCV RNA quantitative is not detectable. Researchers are seeking healthy, pristine cells. Due to the ongoing nature of these chronic viral and bacterial infections, the blood cell populations will change. Researchers want to study changing cell populations as a factor of aging only and not those altered by infections.
5. Ongoing risk factors for HIV or Hepatitis B or C such as: intravenous drug use, non-monogamous unprotected intercourse. These viruses weaken the immune system and cause changes in the white blood cells and their progenitors.
6. Major medical illnesses such as any type of liquid or solid tumor cancer, history of deep vein thrombosis, auto-immune disorders, organ or bone marrow transplant, or liver, kidney, heart or lung disease.
7. A medical finding that shows a participant could not safely go through this procedure. (such as Parkinson s disease, dementia or any uncontrolled behavior that would place the participant s safety at risk)
8. Bleeding conditions such as hemophilia or von Willebrand s disease.
9. Significant abnormalities are found in the results of blood tests such as elevated liver enzymes (2x normal for MedStar Harbor Hospital Clinical Laboratory parameters), abnormal kidney function, positive viral titers, GFR <30.
10. On any medication that can alter blood cell function such as chronic steroid use, antivirals or past or present chemotherapy (complete list located in the Cytapheresis Screening manual stored in the NIA Cytapheresis Unit).
11. Radiation therapy past or present.
12. Inability of researchers to access iliac crest from conditions such as wounds, rashes, or large deposits of adipose tissue that makes localization of the iliac crest difficult.
13. Organ transplant or any graft such as tissue, bone or skin as we don t know how this impacts progenitor cells.

In addition, eligible participants may not be able to participate in a specific bone marrow aspiration procedure but might be eligible at a later date. These include:

1. Pregnancy and Nursing Mothers: Females who are pregnant or who have had a pregnancy in the last 6 weeks are temporarily deferred. They may resume participation in the study 6 weeks after delivery or cessation of lactation and have been cleared by their obstetrician or primary care physician.
2. Medication: Volunteers taking the following medications would be deferred for 2 weeks after course has been completed and volunteer is feeling well: Antibiotics, antifungals, antimalarials.
3. Temporary steroids (tapers): Deferred for 72 hours after symptoms are resolved and prescription is completed if taken orally, intravenously, or intramuscular. No deferral if taken intranasal or for joint injection.
4. Hepatitis B immune globulin: Volunteers are deferred 6 months if given after exposure to hepatitis B to ensure the volunteer has not been infected. If administered for prophylaxis, no deferral is necessary.
5. Live Attenuated Virus Vaccinations: Defer for 4 weeks if symptom-free.
6. Inactivated (Killed Virus) Vaccinations: Defer for 2 weeks if symptom-free.
7. Rabies Vaccine: Deferred for 1 year if given for rabies exposure; otherwise accept immediately if symptom-free.
8. Smallpox Vaccine: Deferred until the scab has separated from the skin spontaneously or 21 days from date of immunization, whichever is longer, if volunteer had no other symptoms or complications. Visual verification of absence of vaccine scab is required. If scab was otherwise removed (not spontaneously separated), defer for 2 months after vaccination date.
9. Experimental Medication or Unlicensed (Experimental) Vaccine is usually associated with a research protocol and the effect on bone marrow is unknown. Deferral is one year unless otherwise indicated by the Principal Investigator.
10. Infection or Fever: Deferred until 2 weeks after antibiotics are completed and volunteer is feeling well.
11. Surgical Procedures: Deferred for 3 months after procedure and released to return to normal activities by primary care physician or surgeon.
12. Close contact with someone else s blood, accidental needle-stick, treatment for syphilis or gonorrhea Volunteers are deferred for 6 months to insure they have not been infected. Viral/serology testing will be repeated and verified as negative prior to bone marrow aspiration procedure.

    1. Received money, drugs or other payment for sex or having sexual contact with a prostitute or anyone else who takes money or drugs or other payment for sex
    2. Has used needles to take drugs, steroids or anything NOT prescribed by their doctor or had sexual contact with anyone who has ever used needles to take drugs or steroids, or anything NOT prescribed by their doctor.
    3. Had sexual contact with or living with anyone who has hepatitis.
    4. Had a tattoo using non-sterile needles or reused ink.
    5. Had a body piercing that used non-sterile needles or multi-use equipment.
13. Had close contact with someone who had a smallpox vaccination such as touching the vaccination site, handling bedding or clothing that has been in contact with an unbandaged vaccination site to insure they have not been infected: Deferral is 2 months if volunteer is symptom-free.
14. Anemia/Leukopenia/Thrombocytopenia:

    1. Volunteers with a hemoglobin of <12.0 for men, <11.0 for women or hematocrit <38 for men, <36 for women may return in 8 weeks to repeat labs to verify anemia. Eligible for procedure once values have returned to normal.
    2. White blood cell count <3.0.
    3. Platelet count <150,000.
    4. Whole blood donation (450 mL) or bone marrow aspiration procedure: Deferred 56 days from date of last donation as mandated by AABB guidelines.
    5. Double unit red cell donation: Deferred for 112 days (16 weeks) as mandated by AABB guidelines.
    6. Platelet or plasma donation: Deferred for 28 days from date of last donation as mandated by AABB guidelines.
    7. There will be no deferral for apheresis donation as we believe it is safe to perform apheresis and bone marrow aspiration on the same day on normal healthy volunteers. For research purposes, we will perform bone marrow aspiration first if both procedures are done on the same day.
15. Received blood transfusion: Deferral is for 12 months to ensure volunteer has not acquired an infectious disease. Annual laboratory testing will be repeated prior to bone marrow aspiration procedure.
16. It is less than six weeks since participation in another research study which is felt by the Principal Investigator to be incompatible with this study. (for example: studies that collect blood, investigational drug studies, vaccine trials, etc.)
17. Travel:

Malaria-endemic countries: Volunteers who are residents of such countries will be deferred for 3 years after departure from the country if they remain free from unexplained symptoms suggestive for malaria. Residence is defined as a continuous stay of longer than 5 years in a country or countries having any malaria-endemic area. Volunteers who are not prior residents of malaria-endemic countries and travel to a malaria-endemic area will be deferred for 12 months after departure from that area. The duration of travel to a malaria-endemic area is defined as more than 24 hours to less than 5 years. Note that a passage greater than 24 hours through a malaria-endemic area while on route to a malaria-free area is considered a sufficient possible exposure to trigger deferral. (A complete list of malarial-endemic countries is kept in the Cytapheresis Screening Manual and is stored in the NIA Apheresis Unit.)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consists of healthy males and females aged 18 years and older. Study subjects are anticipated to be non-patient community volunteers. Individuals will not be excluded based on gender, race or ethnicity. The number of subjects to be enrolled will be 2000. This will allow us to try and maintain 200 active participants.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect bone marrow aspirate for distribution to NIA research investigators for their studies. | Longitudinal study
  We will need to maintain an active volunteer pool of approximately 200 active volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Gupta, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.